CLINICAL TRIAL: NCT04554082
Title: Impact of Zinc to Copper Ratio and Lipocalin 2 in Obese Patients Undergoing Sleeve Gastrectomy.
Brief Title: Evaluation of Micronutrients in Obese Patients
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, hala mourad demerdash, Consultant Clinical Pathology, Alexandria University
Other Study IDs: 0304707; 00018699 (Registry Identifier: FWA); 00012098 (Registry Identifier: IRB)
Record Dates: First submitted 2020-09-06; First posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Nutritional Disorder
Keywords: obesity; zinc; copper; lipocalin 2
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples are stored at -80 for determination of serum copper and zinc and lipocalin 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative Clinical characteristics and metabolic biomarkers: BMI and biochemical parameters including trace elements in patients undergoing laparoscopic sleeve gastrectomy before surgery
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- 9 months' Postoperative metabolic biomarkers: BMI and biochemical parameters including trace elements in patients 9 months after laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — bariatric surgery to loss weight

SUMMARY:
The aim of the study primarily was to investigate the value of zinc to copper ratio as possible biomarker of trace elements imbalance in morbidly obese subjects undergoing LSG.

Secondly to correlate zinc to copper ratio with lipocalin 2 (Lcn2) with respect to Anthropometric measurements and other metabolic biomarkers.

Prospective study will be carried out on 120 morbidly obese adult subjects with a body mass index (BMI) score above 40 along with presence of obesity-related comorbidity. Investigations will be measured preoperative and 9 months postoperative after performing Laparoscopic sleeve gastrectomy; for Body mass index (BMI) and waist circumference. As well as for complete blood count and biochemical biomarkers as fasting blood glucose, lipid profile, serum iron and ferritin. Serum Ceruloplasmin, Zn and Cu levels, followed by calculation of zinc to copper ratio. CRP, serum insulin, serum leptin and lipocalin-2 (Lcn2) will be determined.

DETAILED DESCRIPTION:
CONSORT 2010 Flow Diagram

Materials and methods:

Recruitment Morbidly obese subjects attending clinic at Surgery department for laparoscopic sleeve gastrectomy Alexandria University Hospitals.

Pre-assignment Details adult morbidly obese subjects were included age above 20 years, BMI above 40 Suffering from comorbidities as hypertension, DM, dyslipidemia. Assigned participants were clinically evaluated for comorbidities as hypertension, DM, dyslipidemia.

As well as signs of nutritional deficiency as anemia, brittle nails.

Group Information one group of participants eligible for laparoscopic sleeve gastrectomy were assigned according to their will to participate in study.

Period of evaluation:

First visit: preoperative for clinical assessment of participants, determine BMI and waist circumference and withdrawal of serum blood sample Second visit: within one month after surgery to make sure that no complication occurred after surgery.

Third visit: nine months postoperative for revaluation of participants, determine BMI and waist circumference, and withdrawal of a serum blood sample

Number of participants at initiating the period of study. They were 120 morbidly obese subjects. Number of participants at the end of the period of study. They were 107 subjects, 13 obese subject withdraw from study as they didn't come during follow up period after 9 months.

Participants according Sex (69 females, and 38 male), with the mean age of 41.6±8.9 years. The mean preoperative BMI was 47.43±5.4 kg/m2. Then, they were evaluated 9 months after LSG.

Preoperative and Postoperative Clinical characteristics and metabolic variables in studied subjects.

Preoperative 9 months postoperative P Body weight (Kg) 129.7 ± 12.1 93.4 ±13.6 0.0013* BMI (kg/m2) 47.43±5.4 35.7±3.8 0.0052* Waist circumference (cm) 130.00 ± 4.68 91.82 ± 3.73 0.001* Systolic BP (mmHg) 146.0±17.0 132.0±11.0 0.001* Total cholesterol (mmol/L) 5.85 ± 0.41 4.64 ± 0.31 0.035* Triglycerides (mmol/L) 2.20 ± 0.23 1.92 ± 0.24 0.106 HDL cholesterol (mmol/L) 1.23 ± 0.19 1.39 ± 0.2 0.041* LDL cholesterol (mmol/L) 3.37 ± 0.23 2.97 ± 0.21 0.022* HOMA-IR 2.64 ± 1.3 1.44 ± 0.81 0.013* S. Leptin (ng/ml) 102.87 ± 49.16 33.47 ±12.76 0.0001* CRP (mg/L) 8.4±5.91 3.2±2.98 0.001* Lipocalin 2 (µg/L) 107.24±36.8 51.6±12.73 0.001* Albumin (g/dl) 4.05±0.21 3.91±0.29 0.113

*Statistically significant at (p≤0.05).

Outcome measures:

primarily was to investigate the value of zinc to copper ratio as possible biomarker of TE imbalance in morbidly obese subjects undergoing LSG.

For detection of presence of micronutrient deficiency in morbid obesity in form of zinc to copper ratio and re-evaluate it after loss of weight

Secondly to correlate it with lipocalin 2 (Lcn2) with respect to Anthropometric measurements and other metabolic markers prospectively.

As zinc to copper ratio is considered as biomarker of micronutrient status; therefore, correlate it with other biomarkers of inflammation (lipocalin 2) and other parameters as BMI, FBG to determine if micronutrient status improve after weight loss or not Time frame: 9 months.

Follow-up and outcome parameters:

All studied subjects will be followed up for early postoperative complications (within the first month) as Bleeding or Leak. Then they will be reviewed after 9 months postoperatively for assessment of anthropometric measurements, control of preoperative comorbidities, and manifestations of TE deficiencies (anemia, hair loss, teeth problems, edema. etc.).

Anthropometric parameters

Body mass index (BMI) and waist circumference will be measured preoperative and 9 months postoperative.

Biochemical parameters

Fasting blood samples will be collected from participants prior to surgery and nine months postoperative, after overnight fast and divided into two tubes; EDTA for complete blood count, the rest into plastic tubes and serum sample.

Serum glucose and Total cholesterol, HDL- cholesterol, LDL- cholesterol, and triglyceride, total protein and Albumin. Serum iron (Fe), and ferritin.

Serum insulin, Ceruloplasmin, Zn and Cu levels, CRP and lipocalin-2 (Lcn2) .

Statistical analysis

All data will be analyzed with Statistical Package for the Social Sciences version 20 software (SPSS, Inc., Chicago, IL). Results will be displayed as mean ± SD. Paired Student's t-test used to compare the data pre-operative and nine months postoperative. The chi-squared test used for category variables. Spearman correlation coefficient used to detect the correlation between different variables. Statistical correlations calculated by Pearson's correlation test. P < 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* micronutrient deficiency in morbid obese subjects Adults.
* BMI above 40
* presence of comorbidities as hypertenion, DM, dislipidemia

Exclusion Criteria:

* all causes which might cause micronutrient deficiency as presence of gastroesophageal reflux
* all causes which may cause increase obesity "BMI" as hormonal disturbance ; hypothyroidism or cushing, females receiving contraceptive pills

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult obese subjects with BMI above 40 both males and females presence of obesity comorbidities as hypertension, insulin resistance "type 2 DM" eligible for laporoscopic sleeve gatrectomy
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of zinc to copper ratio as biomarker of micro-nutrient deficiency | nine months
  detect if there are micronutrient deficiency in morbid obesity in form of zinc to copper ratio and re-evaluate it after loss of weight

SECONDARY OUTCOMES:
correlate zinc to copper ratio to lipocalin 2 and other metabolic biomarkers | nine months
  zinc to copper ratio is considered as biomarker of micronutrient status; therefore, it is correlated it with BMI, other biomarkers of inflammation (lipocalin 2) and other parameters as BMI, FBG to determine if micronutrient status improve after weight loss or not

CONTACTS AND LOCATIONS:
Overall Officials: Hala M Demerdash, MD, Principal Investigator — Alexandria University Hospitals

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yerlikaya FH, Toker A, Aribas A. Serum trace elements in obese women with or without diabetes. Indian J Med Res. 2013 Feb;137(2):339-45. PMID 23563378

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04554082/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT04554082/ICF_001.pdf